CLINICAL TRIAL: NCT01109966
Title: A Prospective, Double Blind Randomised Controlled Trial to Evaluate the Immunological Benefits and Clinical Effects of an Elimination Diet Using an Amino Acid Based Formula (AAF)
Brief Title: An Elimination Diet Using a New Amino Acid Based Formula: Immunological and Clinical Effects in Cow's Milk Allergy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CT0140PAICE
Record Dates: First submitted 2010-03-29; First posted 2010-04-23 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Allergy; Food Allergy
Keywords: Allergy; Cow's Milk; Infants; Food Allergy
MeSH Terms: conditions — Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amino acid based formula (Active Comparator): Patients will be randomised to one of two arms:
  Group I: receiving a new amino-acid based formula Group II: receiving a standard AAF formula
  Interventions: Other: Special Medical Food
- New amino acid based formula (Active Comparator): Patients will be randomised to one of two arms:
  Group I: receiving a new amino-acid based formula Group II: receiving a standard AAF formula
  Interventions: Other: Special Medical Food

INTERVENTIONS:
Other: Special Medical Food — Comparison between a standard amino acid based formula and a new amino acid based formula. Subjects with CMA will take their randomised formula for 12 months. Following completion of the intervention (12 months), subjects will transfer to an age appropriate formula and be followed-up at 24 and 36 months.
  Infants should typically consume the following amounts of formula during the study > 500mls/day up to 12 months of age > 400mls/day between 12 and 18 months of age > 300mls/day over 18 months of age.
  Other Names: Amino acid based formula, Neocate LCP
  Arms: Amino acid based formula
Other: Special Medical Food — Comparison between a standard amino acid based formula and a new amino acid based formula. Subjects with CMA will take their randomised formula for 12 months. Following completion of the intervention (12 months), subjects will transfer to an age appropriate formula and be followed-up at 24 and 36 months.
  Infants should typically consume the following amounts of formula during the study > 500mls/day up to 12 months of age > 400mls/day between 12 and 18 months of age > 300mls/day over 18 months of age.
  Other Names: Amino acid based formula
  Arms: New amino acid based formula

SUMMARY:
The purpose of this study is to evaluate whether a new version of an amino acid based formula improves tolerance to milk in cow's milk allergic infants/young children.

DETAILED DESCRIPTION:
Infants with CMA cannot tolerate proteins contained in milk, although they are able to tolerate amino acids which are the 'building blocks' of proteins. Unlike standard infant formulas which are made from milk proteins, amino acid formulas (AAF) are made from nonallergenic aminoacids plus all the other nutrients required to support growth and development.

ELIGIBILITY:
Inclusion Criteria:

* Infants ≤ 8 months of age
* Infants sensitised to cow's milk and diagnosed with IgE mediated cow's milk allergy confirmed by milk challenge or diagnosis of anaphylaxis to milk within the last 3 months

Exclusion Criteria:

* Infants less than 2500 g at birth
* Infants less than 37 weeks gestation
* Infants with severe concurrent illness
* Use of anti- histamines, systemic corticosteroids, systemic antibiotics or anti-mycotic drugs, and immuno-modulatory drugs
* Infants consuming less than 500ml per day of their usual formula at study entry
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study

Max Age: 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the development of oral tolerance in infants with IgE mediated CMA on control or test AAF. | 2 years

SECONDARY OUTCOMES:
To evaluate maturation of the GI immune system in IgE mediated CMA To confirm that the test formula is effective in the dietary management of CMA To assess frequency of other allergies | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Beyer, MD, Principal Investigator — Hospital Charité
Locations (7):
- l'hôpital Necker Enfants malades, Paris, France
- Germany (2):
  - Hospital Charité, Berlin
  - St.-Marien-Hospital, Bonn
- United Kingdom (4):
  - Southampton General Hospital, Southampton, Hampshire
  - David Hyde Allergy Clinic - St. Mary's hospital, Newport, Isle of Wight
  - Evelina Children's Hospital - St Thomas' Hospital, London
  - Newcastle general hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765